CLINICAL TRIAL: NCT06529770
Title: Benefits of Ultrasound-Guided Percutaneous Neuromodulation on the Strength of CrossFit Athletes
Brief Title: Ultrasound-Guided Percutaneous Neuromodulation in the Strength of CrossFit Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Physiotherapist, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMP-e.CF
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy; CrossFit
Keywords: PNM-E; Neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): The group receives no intervention
- NMP-e 3 sessions (Experimental): The group receives 1 session of ultrasound-guided percutaneous neuromodulation. The session wil be received at day 1 of the study.
  Interventions: Other: NMP-e
- NMP-e 1 session (Experimental): The group receives 3 sessions of ultrasound-guided percutaneous neuromodulation. The sessions wil be received at day 1, 7 and 14 of the study.
  Interventions: Other: NMP-e

INTERVENTIONS:
Other: NMP-e — The US-PNM intervention uses a square-wave biphasic current (10 Hz, 250 ms pulse width) at maximum tolerable intensity for 1.5 minutes (10 seconds 10 times), per Fermín Valera and Fran Minaya's protocol. Participants will lie on their side, with the area cleaned and an ultrasound probe cover used.
  Needles (Agu Punt, Spain) will be inserted perpendicularly to target the nerve perineurium. For the axillary nerve (C5-C6), a 0.40/0.50×25 mm needle will be used in a short axis at 80°. For the suprascapular nerve (C5-C6), a 0.30/0.40×25 mm needle will be used.
  Each session involves two needle insertions, with the needle stationary and monitored by a physiotherapist with two years of experience.
  Arms: NMP-e 1 session; NMP-e 3 sessions

SUMMARY:
The origin of CrossFit (CF) dates back to 1995 when Greg Glassman opened the first facility dedicated to the sport he named CF in Santa Cruz, California. However, the dissemination and promotion of this sport began in 2000 with the creation of the CF brand alongside his wife Lauren Jenai. Today, the brand generates around 100 million euros annually and has a market valuation of approximately 4 billion euros. CF boasts 14,000 boxes in 155 countries, with over five million users. Spain ranks as the fifth country with the most CF centers.

CF training focuses on constantly varied functional movements, including gymnastics, weightlifting exercises, and cardiovascular activities (e.g., running or rowing). Variety is one of the main attractions for participants, as the workouts are short, intense, and diverse.

Within invasive physiotherapy, there is the technique of ultrasound-guided percutaneous neuromodulation (US-PNM), which enhances muscle function, muscle recruitment patterns, and motor control. This minimally invasive intervention involves the application of percutaneous electrical stimulation through an electrode similar to an acupuncture needle, placed in close proximity to the nerve or motor point of the target muscle under ultrasound guidance. Performing this technique under ultrasound guidance is recommended as it makes the procedure safer and more effective, allowing real-time visualization of needle positioning and technique application.

Most studies on US-PNM have focused on pain treatment in patients, but some studies have explored its benefits in healthy individuals. For instance, De-la-Cruz-Torre et al. demonstrated that applying this procedure to the sciatic nerve can increase hamstring flexibility; De-la-Cruz-Torres et al. also reported an increase in the performance of the flexor hallucis longus muscle in dancers; Álvarez-Prats et al. showed an improvement in quadriceps muscle strength after performing electrical stimulation on the femoral nerve; and Gallego-Sendarrubias et al. suggested an enhancement in performance skills in soccer players by applying the neuromodulation procedure to the femoral nerve before specific strength training.

Overall, the literature suggests that US-PNM intervention improves strength levels, but the results should be confirmed with future research due to sample size limitations and short-term evaluations. Additionally, there are currently no studies on the application of US-PNM in a sample of CF athletes. Therefore, the objective of this study is to analyze the effectiveness and duration of the effects of two US-PNM protocols applied to the axillary and suprascapular nerves on shoulder rotation strength in healthy CF athletes.

DETAILED DESCRIPTION:
The study aims to:

* Analyze whether 3 sessions of ultrasound-guided percutaneous neuromodulation (US-PNM) are more effective than 1 session of US-PNM for shoulder rotation muscle strength in healthy CrossFit athletes.
* Analyze whether the US-PNM intervention has a positive effect on the ability to perform a one-repetition maximum (1RM) in a functional CF movement, such as the "Shoulder Press," in healthy CrossFit athletes.

To achieve this, a randomized clinical trial is proposed with three study groups:

* Control group: no intervention will be performed.
* Experimental group 1 session US-PNM: will receive 1 session of US-PNM.
* Experimental group 3 sessions US-PNM: will receive 3 sessions of US-PNM, with one week of separation between each session.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old
* Have at least 1 year of experience in CrossFit training

Exclusion Criteria:

* Have not undergone any previous surgeries
* Have no pathology that causes any type of pain
* Have no physical impairment that would hinder dynamometry measurements (muscle injuries, joint instability, joint inflammation, etc.)
* Have no contraindications for the application of Ultrasound-Guided Percutaneous Neuromodulation (US-PNM) such as trypanophobia, pregnancy, epilepsy, or pacemakers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Maximal Strength (1RM) | Measurements will be taken only on the first and last days of the sessions (day 1 and day 21).
  This will be measured using the "shoulder press" exercise.

SECONDARY OUTCOMES:
Internal Shoulder Rotator Muscle Strength. 0º abduction | Measurements will be conducted in all 4 sessions of the study (day 1, day 7, day 13, and day 21).
  Internal shoulder rotation at 0º of shoulder abduction will be measured using dynamometry (Active Force 2), with data collected digitally on the principal investigator's computer.
Internal Shoulder Rotator Muscle Strength. 90º abduction | Measurements will be conducted in all 4 sessions of the study (day 1, day 7, day 13, and day 21).
  Internal shoulder rotation at 90º of shoulder abduction will be measured using dynamometry (Active Force 2), with data collected digitally on the principal investigator's computer.
External Shoulder Rotator Muscle Strength. 0º abduction | Measurements will be conducted in all 4 sessions of the study (day 1, day 7, day 13, and day 21).
  External shoulder rotation at 0º of shoulder abduction will be measured using dynamometry (Active Force 2), with data collected digitally on the principal investigator's computer.
External Shoulder Rotator Muscle Strength. 90º abduction | Measurements will be conducted in all 4 sessions of the study (day 1, day 7, day 13, and day 21).
  External shoulder rotation at 0º of shoulder abduction will be measured using dynamometry (Active Force 2), with data collected digitally on the principal investigator's computer.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, Physiotherapist, Study Director — Universidad de Zaragoza
Locations (2):
- Spain (2):
  - Canvi Crossfit, Tavernes de la Valldigna, Valencia
  - Universidad de Zaragoza, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal

REFERENCES:
- [Derived] Sangiacomo R, Valera-Garrido F, Minaya-Munoz F, Carcasona-Otal A, Herrero P, Lapuente-Hernandez D. Effects of Ultrasound-Guided Percutaneous Neuromodulation on Shoulder Muscle Strength in CrossFit Athletes: A Pilot Randomized Controlled Trial. Neuromodulation. 2025 Jun;28(4):600-610. doi: 10.1016/j.neurom.2025.03.072. Epub 2025 Apr 3. PMID 40183726